CLINICAL TRIAL: NCT04321408
Title: OP2C : Prialt® Observatory in Clinical Practice
Acronym: OP2C
Status: Recruiting | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Esteve (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2019-24
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Refractory Pain
Keywords: Intrathecal analgesia; Ziconotide
MeSH Terms: conditions — Pain, Intractable | interventions — ziconotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ziconotide Injection — Intrathecal analgesia with Ziconotide
  Other Names: Prialt

SUMMARY:
Ziconotide is a strong analgesic marketed since 2005 in Europe and reserved for the intrathecal route. Its efficacy has been proven in particular by 3 randomized clinical studies.

It is particularly effective on neuropathic pain and its main advantages are its power of action, the absence of bone marrow toxicity, and the absence of respiratory depression. In addition, there were no signs of withdrawal when stopping the drug, or of tachyphylaxis.

However, during these studies many adverse reactions were highlighted, especially neuropsychiatric which limited its use. This toxicity was mainly related to the administration of too high doses, especially at the start of treatment (too fast titration).

In recent years, the use of intrathecal ziconotide has become a pertinent option. Indeed, it is recommended as first-line among the intrathecal treatment options.

However, there is a lack of data on the current use of ziconotide in current practice.

The objective of the study will be to describe the practical methods of using intrathecal treatments containing ziconotide.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Severe refractory chronic pain requiring intrathecal analgesia
* Candidate for intrathecal analgesia treatment with ziconotide
* Patient informed about the study and agreeing to take part in.

Exclusion Criteria:

* Contraindications to ziconotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory pain who is initiating treatment with intrathecal analgesia containing ziconotide.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Describe the practical methods of using intrathecal treatments containing ziconotide: indication, initial intrathecal analgesic treatment and evolution of intrathecal analgesic treatment, efficacy and safety in the real clinical practice and monitoring. | 7 years
  Indication, initial intrathecal analgesic treatment and evolution of intrathecal analgesic treatment and monitoring.

SECONDARY OUTCOMES:
Describe the tolerability to intrathecal ziconotide treatment | 7 years
  Tolerability will be assessed by asking questions, clinical examination and paraclinical examinations at each visit
Describe the efficacy on pain of intrathecal ziconotide treatment | 7 years
  The efficacy of the analgesic treatment is measured based on the numeric pain rating scale (0 to 10) at start of Ziconotide, 1, 3, 6, 12 months, and every 12 months thereafter
Estimate the duration of treatment according to the indication | 7 years
  Time between the first and last date of administration of intrathecal ziconotide during study.
Subgroup comparative analysis | 7 years
  Subgroup comparative analysis will be conducted according to initial characteristics, doses course progress of ziconotide and according to efficacy and tolerability.
Responders profile detection | 7 years
  Responders profile according to efficacy on pain of intrathecal ziconotide treatment
Describe quality of life under ziconotide treatment | 7 years
  f) The Quality of life will be assessed by EQ5D-5L questionnaires under intrathecal ziconotide treatment, at 1, 3, 6, 12 months, and every 12 months thereafter until the registry remains open

CONTACTS AND LOCATIONS:
Overall Officials: DENIS DUPOIRON, MD, Study Director — Institut de Canérologie de l'Ouest
Locations (17):
- France (8):
  - Institut de Cancerologie de L'Ouest, Angers
  - Centre Hospitalier Departemental La Roche Sur Yon, La Roche-sur-Yon
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de Montpellier, Montpellier
  - Clinique Breteche, Nantes
  - CHU NICE, Nice
  - Institut Curie, Saint-Cloud
  - Hopital - Foch, Suresnes
- Germany (3):
  - University of Freiburg, Freiburg im Breisgau
  - Justus-Liebig-Universitat, Giessen
  - Jena University Hospital, Jena
- Spain (6):
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital General Universitario Santa Lucía, Cartagena
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Complexo Hospitalario de Ourense, Ourense
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No